CLINICAL TRIAL: NCT03055169
Title: TCF7L2 Polymorphisms Influence on Glycemic Control in ICU Patients With Organ Failure
Acronym: READIAB-G4
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_58; 2010-A00997-32 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-07-13; First posted 2017-02-16 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Genetic Predisposition to Disease; Hyperglycemia; Intensive Care Unit Syndrome; Multiple Organ Failure
Keywords: hyperglycemia; Multiple Organ Failure; biobank; diabetes
MeSH Terms: conditions — Genetic Predisposition to Disease; Hyperglycemia; Multiple Organ Failure; Diabetes Mellitus | interventions — Genetic Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, plasma, mononuclear cells, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intensive care patients: patients with a least one organ dysfunction
  Interventions: Genetic: genetic analysis; Biological: blood and stools samples

INTERVENTIONS:
Genetic: genetic analysis
Biological: blood and stools samples

SUMMARY:
This study evaluates the link between genetic polymorphisms as r7903146, rs12255372 of TCF7L2 gene and the risk of developing hyperglycemia during Intensive care unit stay

ELIGIBILITY:
Inclusion Criteria:

* admission in ICU>48h
* at least one organ dysfunction

Exclusion Criteria:

* age< 18 years
* pregnant women
* admission less than 48h

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in ICU > 48h with at least one organ dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 994 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
value of the odds ratio associated with the relationship between a polymorphism TCF7L2 gene and the occurrence of hyperglycemia | one year after inclusion
  find a link between genetic polymorphism of TCF7L2 and the risk of developing hyperglycemia in intensive care patients with a least one organ dysfunction.
  the hyperglycemia is defined fasting glucose> 1.26 g / l twice or need for treatment with insulin)

SECONDARY OUTCOMES:
Changes in inflammatory markers | one year after inclusion
Changes in serum lipid profile | one year after inclusion
  Changes in cholesterol total, LDL cholesterol, HDL cholesterol and triglycerides
Changes in liver enzymes | one year after inclusion
  Changes in total alanine transaminase (ALT) total gamma-GT total aspartate transaminase (AST)
Insulin Resistance (HOMA) | one year after inclusion
  Calculated using the updated homeostasis model assessment (HOMA) calculator.Higher numbers indicate higher insulin resistance. There are no established cutoffs indicating impaired resistance.

OTHER OUTCOMES:
Blood samples collection | 5 years
  the blood samples collection will created for next research Both on diabetes and / or insulin resistance as its determinisms, at the ICU patient
Number of patients with genotype TCF7L2 by PCR | 5 years
  the prevalence of TCF7L2, in the intensive care patient or not glycemic control, and compared to the values found in the general population.
  the TCF7L2 genes will be evaluated by the Taqman method (7900HT Fast Real-Time PCR System-Applied BioSystem).

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Jourdain, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (5):
- France (5):
  - CHU Cote de Nâcre, Caen
  - Hôpital Roger Salengro, CHRU de Lille, Lille
  - CH Victor Provot, Roubaix
  - CHU Charles Nicolle, Rouen
  - CH Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben Hamou A, Kipnis E, Elbaz A, Bignon A, Nseir S, Tamion F, Du Cheyron D, Jaillette E, Voisin B, Robriquet L, Vanbaelinghem C, Thellier D, Abi Rached H, Jannin A, Duhamel A, Behal H, Machuron F, Espiard S, Preiser JC, Preau S, Pattou F, Jourdain M. Association of transcription factor 7-like 2 gene (TCF7L2) polymorphisms with stress-related hyperglycaemia (SRH) in intensive care and resulting outcomes: The READIAB study. Diabetes Metab. 2020 Jun;46(3):243-247. doi: 10.1016/j.diabet.2019.05.001. Epub 2019 May 20. PMID 31121319